CLINICAL TRIAL: NCT07354113
Title: Feasibility and Acceptability of Peer Intervention for Improving Mental Health Among People Accessing Hormone Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Daphna Stroumsa, Assistant Professor of Obstetrics and Gynecology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00279649; 5K23MD016950-04 (NIH)
Record Dates: First submitted 2026-01-16; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Hormone Care; Mild Depression; Anxiety
Keywords: Peer support group; Enhanced usual care
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Random assignment will be completed using 1:1 computer randomization. Randomization will be stratified by indication and regimen. Randomization will occur prior to the participant's hormone initiation visit to ensure participants assigned to the intervention have standardized access to the peer support components.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Peer support group (Experimental): Participants in the peer support group will be contacted by the peer coordinator to be connected with a peer mentor and will have access to peer support options, namely, one-one one meetings with a peer mentor, group meetings with mentors and other participants, and medical appointment buddy.
  Interventions: Behavioral: Peer support group
- Enhanced Usual Care (EUC) (Other): EUC Documents will be disseminated with hormone care information and resources to share with patients relevant to the participants specific hormone condition or type of hormone care.
  Interventions: Other: Enhanced Usual Care (EUC)

INTERVENTIONS:
Behavioral: Peer support group — A peer mentor will be matched to mentees with participant input. The first meeting is intended to establish contact and expectations. Sessions will be scheduled according to the participant's preferences, with a suggested frequency of once a month with more as necessary and feasible. Participants in the peer support group will have access to peer support options that include: one-one one meetings with a peer mentor; group meetings with mentors and other participants; and medical appointment buddy. Participants are not required to use every option each month. Study visits will be completed baseline-6 months.
  Arms: Peer support group
Other: Enhanced Usual Care (EUC) — Participants randomized to the usual care group will not have access to the peer support options but will complete the study visits (baseline-6 months). All participants will be given a resource document with community resources.
  Arms: Enhanced Usual Care (EUC)

SUMMARY:
The purpose of this study is to test whether the peer support program is acceptable, possible, and can improve mental health among individuals accessing hormone care. Eligible participants will be enrolled and randomized to the support program or enhanced usual care arm. Participants will take part in this study for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hormone condition aged 18 years or older and English speaking
* Initiating or receiving hormone care in Michigan
* Report mild depression or anxiety symptoms, as determined by:

  1. A Patient Health Questionnaire (PHQ9) score ≥ 5 AND/OR
  2. A Generalized Anxiety Disorder (GAD) score ≥ 5.
* Interest or willingness to participate in peer support group meetings either in-person or virtually

Exclusion Criteria:

* Unable to provide informed consent for any reason
* Not fluent in English
* Determination by patient's attending healthcare provider that peer mentorship is not appropriate due to unstable psychosis, cognitive disorder, or severe personality disorder, or other issue
* At imminent risk of suicide, as determined by active suicide ideation with intent and/or a specific plan (endorsed Columbia Suicide Severity Rating Scale number 4 or number 5 in the past month, number 6 in the past 3 months, or spontaneous report)
* Already receiving or intending to receive formalized individual peer specialist services through another community mental health program or organization
* Residing outside of the state of Michigan, or planning to move out of the state of Michigan in the next 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Feasibility assessed by Acceptability based on the average total Abbreviated Acceptability Rating Profile (AARP) score at 6 months | 6 months
  The 9-item AARP is adapted to specifically address this peer support intervention for individuals seeking hormone care. Participants will respond to a 6-point Likert scale rating participants agreement with each acceptability statement. Total scores range from 9-54 with a higher score indicating greater acceptability.
Feasibility based on the number of participants that agreed to participate on the study out of total number of individuals approached for study participation. | Up to 6 months (recruitment period)
Feasibility assessed by Practicality based on the total number of one-on-one in-person sessions vs one-on-one virtual sessions | 6 months
  This is defined as the total number of one-on-one in-person sessions vs one-on-one virtual sessions.
Feasibility assessed by Practicality based on the total the number participants engaged with group sessions in-person vs. number of participants engaged virtually | 6 months
  This is defined as the total number of participants engaged with group sessions in-person vs. number of participants engaged virtually.
Safety based on the number of related adverse events | 6 months
  Related events included will be definitely, probably, and possibly related events (defined per protocol).
  The grading scale that will be used for these events include:
  1. - Mild adverse event (AE) - No treatment needed
  2. - Moderate AE - Resolved with treatment
  3. - Severe AE - Inability to carry on normal activities, required professional medical attention
  4. - Life-threatening or disabling AE
  5. - Fatal AE

CONTACTS AND LOCATIONS:
Overall Officials: Daphna Stroumsa, MD, MPH, MSc, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No